CLINICAL TRIAL: NCT04336735
Title: Improving Immunization Rates in Transplant Candidates Through the Use of a Health Information Technology Tool
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-0527; K08HS026510 (AHRQ)
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Transplantation Infection; Vaccination

STUDY DESIGN:
Intervention Model Description: 45 triads of parents, primary care physicians and subspecialists of children awaiting heart, liver and kidney transplantation will be enrolled to use a novel immunization tool (app).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunization Tool Users (Experimental): Users will trial a novel transplant-specific immunization tool (app)
  Interventions: Other: immunization app

INTERVENTIONS:
Other: immunization app — A transplant specific immunization app will be trialed that 1) provides vaccine information and education, 2) stores vaccine records and 3) provides reminders when vaccines are due

SUMMARY:
Vaccine preventable infections are a serious complication following pediatric solid organ transplant. Immunizations are a minimally invasive and cost-effective was to reduce these infections. Despite the importance of pre-transplant vaccination, the majority of pediatric solid organ transplant recipients are not up-to-date on age-appropriate immunizations at the time of transplant. The goal of this study is to pilot a novel health information technology immunization tool to improve immunization rates in pediatric solid organ transplant candidates.

DETAILED DESCRIPTION:
Triads of parents, primary care physicians, and transplant sub-specialists will be enrolled to use a pre-transplant immunization tool while their child awaits transplant. The tool will provide information about vaccines, information about vaccine-preventable infections in the transplant population, a central easily accessible vaccine record, and a communication portal. The tool will also send vaccine reminders when vaccinations are due. The investigators will assess 1) the effectiveness of the tool in improving pre-transplant immunization rates, 2) the acceptability of the tool to users and 3) the feasibility of the tool.

ELIGIBILITY:
Inclusion Criteria:

* Parent, primary care provider and sub-specialist of a child awaiting heart, liver or kidney transplant

Exclusion Criteria:

* Non English speaking
* No access to a smart phone or computer

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Transplant Immunization Tool, as measured by number of patients with up-to-date vaccinations | Date of transplantation (up to 3 years post-enrollment)
  We will assess whether the novel immunization tool improves pre-transplant vaccination rates. The number of participants who are up to date with vaccinations will be reported.

SECONDARY OUTCOMES:
Acceptability and Feasibility of the Transplant Immunization Tool, as assessed by a questionnaire | Date of transplantation (up to 3 years post-enrollment)
  We will assess whether the novel immunization tool is feasible and acceptable to users using a Likert scale with possible scores of 1-5, with 1 being least feasible/acceptable to the participant and 5 being the most feasible/acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Feldman, Principal Investigator — UCD
Locations (1):
- Childrens Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No